PRINCIPAL INVESTIGATOR: Jing Wu, MD, PhD

STUDY TITLE: Phase II trial evaluating Nivolumab in patients with recurrent IDH-mutant

gliomas with and without hypermutator phenotype

STUDY SITE: NIH Clinical Center

Cohort: Standard

Consent Version: 10/30/2024

# WHO DO YOU CONTACT ABOUT THIS STUDY?

Principal Investigator: Jing Wu, MD, PhD

Email: jing.wu3@nih.gov

Ph: 240-760-6036

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers. Taking part in research at the NIH is your choice.

If the individual being asked to participate in this research study is not able to give consent to be in this study, you are being asked to give permission for this person as their decision-maker. The term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research, throughout the remainder of this document.

## IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

## WHY IS THIS STUDY BEING DONE?

The purpose of this study is to determine whether the experimental drug, nivolumab can increase the time it takes for your disease to get worse.

Nivolumab has been approved by the U.S. Food and Drug Administration (FDA) for patients with some types of cancers, but not glioma. Therefore, nivolumab is considered experimental in this study.

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 10/30/2024




Nivolumab has already been tried in other studies to treat people with glioma and was shown to be safe.

Nivolumab is an agent that targets and blocks a pathway that prevents your immune system from effectively fighting your cancer.

Gliomas are the most common malignant brain tumors. Gliomas are classified by location, grade, clinical and molecular features. One of the molecular features includes specific changes (mutations) in the genes IDH1 or IDH2. Another molecular feature is total amount of mutations in the tumor, which can be high and called hypermutator phenotype (HMP) or low and called non-hypermutator phenotype (NHMP). We believe that nivolumab can be more effective in patients with IDH1 or IDH2 mutated gliomas with the hypermutator phenotype, but we do not know for sure. Considering this, we will enroll people with IDH1 or IDH2 mutated gliomas with and without HMP.

#### WHY ARE YOU BEING ASKED TO TAKE PART IN THIS STUDY?

You are being asked to be part of this study because you have been diagnosed with glioma that has specific changes (mutations) in genes IDH1 or IDH2.

# HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

Up to 70 people will be enrolled on the study, but because not everyone will be eligible, it is expected that 59 will be treated.

## **DESCRIPTION OF RESEARCH STUDY**

# **During the study**

If it is determined that you are eligible for the study, nivolumab will be administered to you by IV (through an intravenous catheter, a small plastic tube that is put into a vein, usually in your arm) on days 1 and 15 of the first 2 cycles and then only on day 1 of the following cycles 3-16 (1 Cycle = 4 weeks).

You will continue treatment with nivolumab until your disease gets worse, you have unacceptable side effects, or you have completed 16 months of study therapy, whichever comes first.

Treatment and all study involved procedures will be done during outpatient visits.

Before treatment starts, you will have an electrocardiogram (EKG – a record of your heartbeat) to evaluate your heart.

Ongoing Procedures before treatment on the day 1 of each cycle

- Physical examination, including weight, neurologic assessment and vital signs. Vital signs will be taken on the days you receive nivolumab.
- Review of your symptoms, medications and your ability to perform your normal activities.
- Routine blood tests (about 2 teaspoons) to find out if you are anemic, have low blood counts, and if your liver, kidneys, and other organs are working well.

Additional Procedures before treatment on first day of each cycle:

• Pregnancy test if you are a woman who can have children.

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




• Imaging Assessments – MRI of brain every 8 weeks. An MRI creates pictures of your brain using strong magnets instead of x-ray energy. At the time of each scan, you will be asked to fill out a screening form to verify that it is safe for you to have the scan. You will also be asked to remove any metallic objects you may be wearing (for example, watches, earrings or piercings) and possibly to change into a hospital gown. Then you'll be asked to lie on a narrow bed that will move into the MRI scanner. Once you are comfortable, the table will be moved into the scanner (the scanner is a long, narrow tube that is open at each end). You will need to lie still on the table during the scan which will take about 30 -45 minutes to complete. You will hear normal "hammering" or clicking and squealing noises during the scan. While in the scanner you will be fitted with earplugs or earmuffs to muffle the sound. You will be able to communicate with the technician running the scan the entire time and will be provided an emergency button to squeeze at any time if you decide you want the scan to stop.

#### Research tests

In addition to the tests that we will conduct to determine whether you are having side effects or if you are responding to the study therapy, and the genetic testing on blood or saliva performed at screening, we will also collect additional samples from you for purposes of research only. These studies include:

- Blood samples before initiation of treatment and every month for the first 3 months. The amount of blood taken is about 12 teaspoons. Every other month thereafter, and when your disease progresses the amount taken is about 9 teaspoons. These samples will study how well your immune system fights the tumor.
- Collecting of tumor samples from surgery/biopsy to study molecular markers of your tumor, all genes in your tumor, how efficiently they are working, genetic changes that can be connected to tumor development and response to treatment.
- You will be asked to complete a questionnaire to determine your general well-being and function before the start of the treatment and approximately every 8 weeks after that (before imaging studies). It will take you about 5 minutes and will only be done if you can complete the surveys in English.

# Tumor Collection (at Progression)

If your tumor progresses while you are on the study and you need to undergo surgery, if you agree, we would like to collect a portion of the tumor so we can evaluate it for tumor markers. The research that may be done with your tissue at progression is not designed specifically to help you. It might help people who have cancer in the future.

## Genetic testing and return of results

Your samples contain genes, which are made up of DNA (deoxyribonucleic acid) which serves as the "instruction book" for the cells that make up our bodies. We will use the tissue samples and blood you provided to learn about how the genes in your tumor compare to genes in normal tissue. Your tissue will help us study how genes might play a role in rare cancer and other diseases. We will not share the results of these research tests with you.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




When we are conducting the above genetic tests, it is possible that we could identify changes in other parts of your DNA that are not related to this research. These are known as "incidental medical findings":

- Changes in genes that are related to diseases other than cancer
- Changes in genes that are not known to cause any disease. These are known as normal variations.
- Changes in genes that are new and of uncertain clinical importance. This means that we do not know if they could cause or contribute to a disease or if they are normal variations.

However, the analyses that we perform in our laboratory are for research purposes only; they are not nearly as sensitive as the tests that are performed in a laboratory that is certified to perform genetic testing. Changes that we observe unrelated to our research may or may not be valid. Therefore, we do not plan to inform you of the results of testing on your tissue and blood that is performed in our research lab. However, in the unlikely event that we discover a finding that is believed to be clinically important based on medical standards at the time that we first analyze your results, we will contact you. This could be many years in the future. We will ask you to have an additional tube of blood drawn to verify the findings we have seen in our lab. If the results are verified, you will be re-contacted and offered a referral to a genetic healthcare provider to discuss the results.

You should not assume that if you are not contacted, you do not have any gene variants that might be related to a disease.

# When you are finished taking the drugs

Approximately 28, 60 and 100 days after you have finished taking the study drug, you will be asked to return to Clinical Center for a safety follow up visits. At these visits, your will be asked questions about your health, get a physical and neurological exam, undergo blood tests, and might have an MRI of your brain.

If you still have unresolved health issues, caused by study drug, you will be invited to NIH for additional tests and treatment.

If your disease did not get worse, but you finished taking nivolumab before 1 year of getting treatment, we will invite you for imaging studies approximately every 8 weeks. These visits will continue until 1 year from beginning of treatment or until your disease get worse, whatever comes first.

If you are unable to return for these visits, we will obtain the information from you by telephone or e-mail.

After these safety visits we will call or e-mail you every 6 months to ask you to complete questionnaires to determine your general well-being and function. These questionnaires can be completed electronically, so you do not need to come to Clinical Center for this.

## **BIRTH CONTROL**

If you are a woman who is breast feeding or pregnant, you will not take part in the study because we don't know how this medicine would affect your baby or your unborn child. If you are a woman

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




who can become pregnant, you will need to practice an effective form of birth control before starting study treatment, during study treatment and for 5 months after the last drug infusion. If you think that you are pregnant, you should tell your study doctor or nurse at once.

Effective forms of birth control include:

- abstinence
- intrauterine device (IUD)
- hormonal [birth control pills, injections, or implants]
- Barrier method of birth control: condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide
- tubal ligation
- partner's vasectomy

## RISKS OR DISCOMFORTS OF PARTICIPATION

# What side effects or risks can I expect from being in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work or home and spend more time in the hospital or doctor's office than usual
- You may be asked sensitive or private questions which you normally do not discuss

Nivolumab used in this study may affect how different parts of your body work such as your liver, kidneys, heart, blood and brain. The study doctor will be testing your blood and perform neurological exam and will let you know if changes occur that may affect your health.

Here are important points about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.
- Some side effects may interfere with your ability to have children.
- Some side effects may be serious and may even result in death.

Here are important points about how you and the study doctor can make side effects less of a problem:

- Tell the study doctor if you notice or feel anything different so they can see if you are having any symptoms.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce side effects.
- Late side effects of the investigational agents may affect your ability to tolerate subsequent regimens of standard of care chemotherapy.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




Below we show the most common and the most serious side effects that researchers know about. There might be other side effects that researchers do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

## Risks from Nivolumab

Side effects of nivolumab may happen anytime during treatment or even after your treatment has ended. Some of the common and less common side effects can be serious. Call or see your healthcare provider right away if you develop any problems listed below or if the symptoms get worse.

## **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving nivolumab, more than 20 and up to 100 may have:

Tiredness

## OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving nivolumab, from 4 to 20 may have:

- Rash, itching
- Anemia which may require blood transfusion
- Swelling and redness of the eye
- Pain
- Diarrhea, nausea
- Dry mouth
- Fever
- Swelling and redness at the site of the medication injection
- Bruising, bleeding
- Pain or swelling of the joints
- Loss of appetite
- Reaction during or following a drug infusion which may cause fever, chills, rash
- Nivolumab may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:
  - o Lung problems (pneumonitis and pleural effusion). Symptoms may include: new or worsening cough, chest pain, shortness of breath.
  - Intestinal problems (colitis) that can rarely lead to tears or holes in your intestine.
     Signs and symptoms of colitis may include: diarrhea or increase in bowel movements, blood in your stools or dark, tarry, sticky stools, severe belly pain or tenderness.
  - O Skin: itching; rash, blisters including inside the mouth; loss of skin pigment
  - o Liver problems (hepatitis) which can cause liver failure. Signs and symptoms of hepatitis may include: yellowing of your skin or the whites of your eyes, severe

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




- nausea or vomiting; drowsiness; pain in the right upper belly
- O Hormone gland problems (especially the thyroid, pituitary and adrenal glands, and pancreas). Signs and symptoms may include: headaches that will not go away or unusual headaches, extreme tiredness or changes in mood or behavior; decreased sex drive; weight loss or weight gain; excessive thirst or urine; dizziness or fainting.

# RARE, AND SERIOUS

In 100 people receiving nivolumab, 3 or fewer may have:

- Dry eyes
- Eye pain, eyelid swelling and redness, restricted or limited eye movement
- Sores in the mouth which may cause difficulty swallowing
- Nivolumab may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:
  - Visual disturbances which may cause double vision, blurred vision, or loss of vision with a chance of blindness
  - A condition with high blood sugar which leads to tiredness, frequent urination, excessive thirst, headache, nausea and vomiting, and can result in coma
  - Kidney problems, including nephritis and kidney failure requiring dialysis. Signs
    of kidney problems may include: decrease in the amount of urine, blood in your
    urine, ankle swelling.
  - Heart problems including swelling and heart failure. Symptoms and signs of heart problem may include: Shortness of breath, swelling of the ankle and body.
  - o Problems with the stomach that can lead to symptoms like stomach pain, cramping, diarrhea, nausea and vomiting.
  - o Problem of the muscle, including swelling, which can cause muscle pain and severe muscle weakness sometimes with dark urine
  - Swelling of the brain (meningitis/encephalitis) which may cause: headache, stiff neck, confusion, sleepiness, seizures or injury to the brain which may cause headache, seizure, blindness (also known as Reversible Posterior Leukoencephalopathy Syndrome)
  - Problem of the nerves that can cause paralysis. Signs and symptoms may include: numbness, tingling of hands and feet; weakness of the arms, legs and facial muscle movement
  - Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
  - Complications associated with stem cell transplant using donor stem cells (allogeneic stem cell transplant). These complications are caused by attack of donor cells on the host organs (inducing liver, skin and gut damage), and can lead

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




to death. If you are considering an allogeneic stem transplant after participating in this study, please tell your doctor that you have received nivolumab therapy, since the risk and severity of transplant-associated complications may be increased.

Getting medical treatment right away may keep these problems from becoming more serious. Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

# Risks for gadolinium enhanced MRI scans:

## **Procedure**

People are at risk for injury from the MRI magnet if they have some kinds of metal in their body. It may be unsafe for you to have an MRI scan if you have pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metal prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, tattoos, an implanted delivery pump, or shrapnel fragments. Welders and metal workers may have small metal fragments in the eye. You will be screened for these conditions before having any MRI scan. If you have a question about metal in your body, you should inform the staff. You will be asked to complete an MRI screening form before each MRI scan you have.

In addition, all magnetic objects (like watches, coins, jewelry, and credit cards) must be removed before entering the MRI scan room.

People with fear of confined spaces may become anxious during an MRI. Those with back problems may have back pain or discomfort from lying in the scanner. The noise from the scanner is loud enough to damage hearing, especially in people who already have hearing loss. Everyone having a research MRI scan will be fitted with hearing protection. If the hearing protection comes loose during the scan, you should let us know right away.

There are no known long-term risks of MRI scans.

During part of the MRI you will receive gadolinium, a contrast agent, through an intravenous (iv) catheter. It will be done for medical purposes.

It is not known if MRI with contrast is completely safe for a developing fetus. Therefore, all women of childbearing potential will have a pregnancy test performed no more than 24 hours before each MRI scan with contrast. The scan will not be done if the pregnancy test is positive.

#### Risks

The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000 people, more severe symptoms have been reported including shortness of breath, wheezing, hives,

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis (NSF)". This condition always involves the skin and can also involve the muscles, joints and internal organs. NSF has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is below the safe level.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA has issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The long-term effects of the retained gadolinium are unknown. Some types of gadolinium contrast drugs are less likely to remain in the body than others. We use gadobutrol which is a form of gadolinium contrast that is less likely to accumulate in the body than older types of gadolinium. You will receive additional information called a medication guide about the contrast medication you will receive.

Please tell your research team if you have had any MRI scans in the past 12 months. We will also give you additional information called a "Medication Guide." Upon request, we will give you individual information about retained gadolinium we see on your studies.

# Risks of Electrocardiograms

Skin irritation or discomfort may occur at the site where the ECG electrodes (sticky patches) are taped to your skin. The test is painless and takes less than a minute to perform. After the test, the electrodes are removed.

# **Risks from Blood Collection**

Side effects of blood draws include pain and bruising in the area where the needle was placed, lightheadedness, and rarely, fainting. When large amounts of blood are collected, low red blood cell count (anemia) can develop.

## **Risks from Questionnaires**

Questionnaires contain questions that can be sensitive for you to answer.

## **Privacy Risks**

The following general points are indirectly related to your participation in the research study.

Privacy Risks Associated with Genetic Testing

It may be possible that genetic information from you could be used by law enforcement agencies or other entities to identify you or your blood relatives.

Psychological or Social Risks Associated with Return of Incidental or Secondary Findings

As part of the research study, it is possible that you could learn that you have genetic risks for another disease or disability. This may be upsetting and, depending on what you learn, might create a need to make challenging decisions about how to respond.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




Although your genomic information is unique to you, you share some genomic similarities with your children, parents, brothers, sisters, and other blood relatives. Therefore, learning your research results could mean something about your family members and might cause you or your family distress. Before joining the study, it may be beneficial to talk with your family members about whether and how they want you to share your results with them.

Protections against misuse of genetic information

This study involves genetic testing on samples. Some genetic information can help predict future health problems of you and your family and this information might be of interest to your employers or insurers. The Genetic Information Nondiscrimination Act (GINA) is a federal law that prohibits plans and health insurers from requesting genetic information or using genetic information. It also prohibits employment discrimination based on your health information. However, GINA does not address discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA also does not protect you against discrimination based on an already-diagnosed condition or disease that has a genetic component.

## POTENTIAL BENEFITS OF PARTICIPATION

# Are there benefits to taking part in this study?

The aim of this study is to find out whether the experimental treatment can increase the time it takes for your disease to get worse. We do not know if you will receive personal, medical benefit from taking part in this study. Potential benefits could include shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer. Because there is not much information about the drug's effect on your cancer, we do not know if you will benefit from taking part in this study, although the knowledge gained from this study may help others in the future who have cancer.

## ALTERNATIVE APPROACHES OR TREATMENTS

Instead of being in this study, you have these options:

- Getting standard FDA approved treatment or care for your cancer without being in a study
- Taking part in another study
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Please talk to your doctor about these and other options.

# STOPPING THERAPY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease comes back during treatment
- if you need to take medication that is not allowed on the study

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




- if you become pregnant
- if you have side effects from the treatment that your doctor thinks are too severe
- if new information shows that another treatment would be better for you
- if the investigator decides to end the study

In this case, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to Bristol-Myers Squibb or designated representatives. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases cannot be recalled and destroyed.

# **CONFLICT OF INTEREST (COI)**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

Bristol-Myers Squibb is providing nivolumab for this study to NIH without charge. No NIH employee involved in this study receives any payment or other benefits from Bristol-Myers Squibb.

#### USE OF SPECIMENS AND DATA FOR FUTURE RESEARCH

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

These specimens and data will be used for future research and shared with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

We may put your research data in a large database for broad sharing with the research community. These databases are commonly called data repositories. These data repositories might or might not

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




be located at the NIH. The information in this database could include but is not limited to genetic information, ethnicity and sex. If your individual research data is placed in one of these repositories, it will not be labeled with your name or other information that could be used to easily identify you, and only qualified researchers will be able to look at your data. These researchers must receive prior approval from individuals or committees to access the data. Your summary genomic data is being placed *in an* unrestricted database, so researchers will be able to access summary information about all the participants included in the study (including you), or summary information combined from multiple studies, without applying for permission. The risk of anyone identifying you with this information is very low.

If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

# **Genomic Data Sharing**

As part of this research study, we will put your genomic data in a large database for broad sharing with the research community. These databases are commonly called data repositories. The information in this database will include but is not limited to genetic information, race and ethnicity, and sex. If your individual data are placed in one of these repositories, they will be labeled with a code and not with your name or other information that could be used to easily identify you, and only qualified researchers will be able to access them. These researchers must receive prior approval from individuals or committees with authority to determine whether these researchers can access the data.

Summary information about all of the participants included in this study (including you) is being placed in a database and will be available through open access. That means that researchers and non-researchers will be able to access summary information about all the participants included in the study, or summary information combined from multiple studies, without applying for permission. The risk of anyone identifying you with this information is very low.

NIH policies require that genomic data be placed in a repository for sharing. Therefore, we cannot offer you a choice of whether your data will be shared. If you do not wish to have your data placed in a repository, you should not enroll in this study.

## COMPENSATION, REIMBURSEMENT, AND PAYMENT

# Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this study.

# Will you receive reimbursement or direct payment by NIH as part of your participation?

On this study, the NCI will reimburse the cost for some of your expenses such as those for hotel, travel, meals. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. The amount and form of these payments are determined by the NCI Travel

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




and Lodging Reimbursement Policy. You will be given a summary of the policy which provides more information.

If your travel to the NIH Clinical Center (e.g. flight, hotel) is arranged and paid for by the NIH, the agency making the reservations and their representatives will have access to your identifiable information.

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

# CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor, Center for Cancer Research, NCI, or their agents
- Qualified representatives from Bristol-Myers Squibb, the pharmaceutical company who produces nivolumab.

The researchers conducting this study and the NIH follow applicable laws and policies to keep your identifying information private to the extent possible. However, there is always a chance that, despite our best efforts, your identity and/or information about your participation in this research may be inadvertently released or improperly accessed by unauthorized persons.

In most cases, the NIH will not release any identifiable information collected about you without your written permission. However, your information may be shared as described in the section of this document on sharing of specimens and data, and as further outlined in the following sections.

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

# **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

## **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical records we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

# POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




# PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Jing Wu, M.D., PhD, Email: jing.wu3@nih.gov Telephone: 240-760-6036. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

# **CONSENT DOCUMENT**

Please keep a copy of this document in case you want to read it again.

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




| Signature of Research Participant | Print Name of Research Particip | pant Date |
|---|---|---|
| about this study and have been gi<br>authorized to make research decision<br>authority to provide consent to this s | e (LAR) for an Adult Unable to Consent: ven the opportunity to discuss it and to a cons on behalf of the adult participant unable tudy. As applicable, the information in the abusent who agrees to participate in the study. | sk questions. I am lega<br>le to consent and have |
| Signature of LAR | Print Name of LAR | Date |
| Investigator: | | |
| <del>_</del> | Print Name of Investigator r: ess has been used to enroll a non-English e full consent has been used to enroll a blir | |
| Witness should sign below if either 1. A short-form consent proc | r:<br>ess has been used to enroll a non-English | speaking subject or |
| Witness should sign below if either 1. A short-form consent proc 2. An oral presentation of the | r:<br>ess has been used to enroll a non-English | speaking subject or |
| Witness should sign below if either 1. A short-form consent proc 2. An oral presentation of the Witness: Signature of Witness* | r:<br>ess has been used to enroll a non-English<br>e full consent has been used to enroll a blin | speaking subject or nd or illiterate subject Date |
| Witness should sign below if either 1. A short-form consent proc 2. An oral presentation of the Witness: Signature of Witness* *NIH ADMINISTRATIVE SECTINTERPRETER: | r: ess has been used to enroll a non-English e full consent has been used to enroll a blin Print Name of Witness | speaking subject or nd or illiterate subject Date DING THE USE OF |
| Witness should sign below if either 1. A short-form consent proce 2. An oral presentation of the Witness: Signature of Witness* *NIH ADMINISTRATIVE SECTINTERPRETER: An interpreter, or other indiverse facilitated | r: ess has been used to enroll a non-English e full consent has been used to enroll a bline a print Name of Witness TION TO BE COMPLETED REGARD | speaking subject or and or illiterate subject Date Ding The USE OF An angular preferred language. |
| Witness should sign below if either 1. A short-form consent proce 2. An oral presentation of the Witness: Signature of Witness* *NIH ADMINISTRATIVE SECTINTERPRETER: An interpreter, or other individual facilitated the administration of informed consulso serve as the witness. | r: ess has been used to enroll a non-English e full consent has been used to enroll a blind a blind print Name of Witness FION TO BE COMPLETED REGARD idual, who speaks English and the particular particular idual. | Date Date Ding THE USE OF A spant's preferred languate obtaining consent may |


IRB NUMBER: 19C0006 IRB EFFECTIVE DATE: 11/4/2024

| MEDICAL RECORD | CONSENT TO PARTICIPATE IN AN NIH CLINICAL RESEARCH STUDY |
|---|---|
| providing interpretive support | is: |

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1) Version Date: 10/30/2024


